CLINICAL TRIAL: NCT02814890
Title: Thoracic Paravertebral Block Using Ropivacaine With/Without Dexmedetomidine in Video-assisted Pneumonectomy
Brief Title: Thoracic Paravertebral Block Using Ropivacaine and Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianghui Xu (Other)
Responsible Party: Sponsor-Investigator, Jianghui Xu, MD, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011QD10
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
Keywords: Thoracic paravertebral block; Dexmedetomidine; Video-assisted Pneumonectomy; Ropivacaine; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine and dexmedetomidine (Experimental): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine + 1μg/kg dexmedetomidine at the end of video-assisted pneumonectomy.
  Interventions: Procedure: Video-assisted Pneumonectomy; Procedure: Thoracic paravertebral block
- Ropivacaine only (Active Comparator): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine at the end of video-assisted pneumonectomy.
  Interventions: Procedure: Video-assisted Pneumonectomy; Procedure: Thoracic paravertebral block

INTERVENTIONS:
Procedure: Video-assisted Pneumonectomy — Video-assisted Pneumonectomy under general anesthesia.
Procedure: Thoracic paravertebral block — The procedure is guided by ultrasound combined with nerve stimulator at T3-4, T4-5, T5-6, T6-7 of surgical side.
  Other Names: Thoracic paravertebral nerve block

SUMMARY:
The hypothesis of the study is whether dexmedetomidine plus local anesthetic ropivacaine could extend the pain relieve time compared with only ropivacaine when thoracic paravertebral block is performed at the end of video-assisted pneumonectomy.

DETAILED DESCRIPTION:
The investigators aim to recruit 60 patients undergoing video-assisted pneumonectomy. All patients ASA physical status I-II grade, aged within 20-70 years, are randomly allocated into two groups: 75mg/20ml ropivacaine only group (Group R, n=30) and 75mg/20ml ropivacaine + 1μg/kg dexmedetomidine (Group RD, n=30). At the end of surgery, the investigators perform four points thoracic paravertebral block guided by ultrasound combined with nerve stimulator at T3-4, T4-5, T5-6, T6-7 of surgical side where 5ml solution is injected to each point. The characteristics of patients are analyzed to confirm whether they are comparable in both groups. Pain was assessed according to a numerical rating scale (NRS) (0 = no pain; 10 = worst pain imaginable). Patients were asked to evaluate the maximal degree of pain. Pain scores were recorded in post anesthesia care unit(PACU), and1, 2,4, 8, 12, 24, 36 and 48 hours after surgery. The study endpoints are evaluated by an anesthesiologist who does not know the group allocation. The postoperative rescue analgesic administration, adverse outcomes and patient satisfaction are also recorded.

All data were processed in SPSS 18.0 (SPSS Inc., Chicago, IL USA). Normality was tested by the Kolmogorov-Smirnov analysis. Comparisons of continuous outcomes among groups were examined using Kruskal-Wallis test. Chi-square analysis or Fisher's exact test was used to assess categorical outcomes between groups. A P-value<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II grade
* Undergoing elective video-assisted pneumonectomy under general anesthesia.
* Participants aged from 30-70 years old.

Exclusion Criteria:

* Refusal for paravertebral block
* Inability to obtain informed consent
* Coagulation disorders, neuropathy, or body mass index greater than 40 kg/m2
* Pregnancy
* Infections at the site of injection for the paravertebral block
* Allergy to local anesthetics or alpha-2 adrenergic agonists
* Heart block or bradycardia (heart rate < 60 beat per minute)
* Clinically significant cardiovascular, pulmonary, renal, or hepatic diseases

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD,PhD, Study Chair — Department of Anesthesiology,Huashan Hospital,Fudan University
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-five patients were initially recruited in Auguest, 2016.
Pre-assignment Details: The participants who were converted to thoracotomy because of intraoperative bleeding or pleural adhesions would be wash out.
Groups:
- Group RD(Ropivacaine and Dexmedetomidine): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine + 1μg/kg dexmedetomidine at the end of video-assisted pneumonectomy.
  Video-assisted Pneumonectomy: Video-assisted Pneumonectomy under general anesthesia.
  Thoracic paravertebral block: The procedure is guided by ultrasound combined with nerve stimulator at T4-5, T5-6, T6-7, T7-8 of surgical side.
  Sixty-five patients were initially recruited. Five patients were excluded from present study, including 3 patients in group RD who were converted to thoracotomy because of intraoperative bleeding or pleural adhesions.
- Group R(Ropivacaine Only): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine at the end of video-assisted pneumonectomy.
  Video-assisted Pneumonectomy: Video-assisted Pneumonectomy under general anesthesia.
  Thoracic paravertebral block: The procedure is guided by ultrasound combined with nerve stimulator at T4-5, T5-6, T6-7, T7-8 of surgical side.
  Sixty-five patients were initially recruited. Five patients were excluded from present study, including 2 patients in group R who were converted to thoracotomy because of intraoperative bleeding or pleural adhesions.
Period: Overall Study
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Started | 33 | 32
Completed | 30 | 30
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group RD(Ropivacaine and Dexmedetomidine): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine + 1μg/kg dexmedetomidine at the end of video-assisted pneumonectomy.
  Video-assisted Pneumonectomy: Video-assisted Pneumonectomy under general anesthesia.
  Thoracic paravertebral block: The procedure is guided by ultrasound combined with nerve stimulator at T4-5, T5-6, T6-7, T7-8 of surgical side.
  There were no significant differences between two groups in demographic and operative data(Gender, Age, Weight, Height, ASA（Ⅰ/Ⅱ), FEV1 (% predicted), FEV1/FVC (% predicted), Intraoperative fentanyl, Duration of surgery, Duration of anesthesia).
- Group R(Ropivacaine Only): Thoracic paravertebral block is performed using 75mg/20ml ropivacaine at the end of video-assisted pneumonectomy.
  Video-assisted Pneumonectomy: Video-assisted Pneumonectomy under general anesthesia.
  Thoracic paravertebral block: The procedure is guided by ultrasound combined with nerve stimulator at T4-5, T5-6, T6-7, T7-8 of surgical side.
  There were no significant differences between two groups in demographic and operative data(Gender, Age, Weight, Height, ASA（Ⅰ/Ⅱ), FEV1 (% predicted), FEV1/FVC (% predicted), Intraoperative fentanyl, Duration of surgery, Duration of anesthesia).
- Total: Total of all reporting groups
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only) | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: 5 patients were excluded due to their type of surgery transfering from VATS to thoracotomy, in which 3 patients in Group RD and 2 ones in Group R.
  years
    recruited number of participants | 59.2 (9.6) | 59.7 (9.4) | 59.6 (9.3)
    analyzed number of participants: number analyzed (Participants) | 30 | 30 | 60
    analyzed number of participants | 59.2 (9.7) | 59.5 (9.7) | 59.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 patients were excluded due to their type of surgery transfering from VATS to thoracotomy, in which 3 patients in Group RD and 2 ones in Group R.
  Participants
    number analyzed (Participants) | 30 | 30 | 60
    Female | 12 | 13 | 25
    Male | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain (Pain Scores) Intensity Measure
Description: Pain Numerical Rating Scales （NRS) at rest（0: no pain--means the minimum value; 10: worst possible pain--means the maximum value)
Time Frame: assessed over 48 hours after surgery, self reported pain intensity at 2 days reported
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Group RD(Ropivacaine and Dexmedetomidine); Group R(Ropivacaine Only): The pain scores (numerical rating scale, NRS) postoperative 48h at rest and coughing were assessed.
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Number analyzed (Participants) | 30 | 30
units on a scale | 1 [0 to 2] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Group RD(Ropivacaine and Dexmedetomidine) vs Group R(Ropivacaine Only); Sample size: Based on our previous data, pain score at rest 48 hours postoperatively when using ropivacaine only was of 2.8 with a standard deviation of 1.4. Assuming a decrease of pain score by 1.1 being clinically significant, twenty six patents in each group would be required for a study power of 80% (α=0.05,β=0.2). Considering possible dropouts, we aimed at recruiting 30 patients in each group with a total of 60 patients; Test type: Other — difference test; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Patient Satisfaction
Description: using a 5-point Likert scale (5-point: completely satisfied, 4-point: quite satisfied, 3-point: slightly dissatisfied, 2-point: dissatisfied, 1-point: very dissatisfied)
Time Frame: Hour 48 after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Group RD(Ropivacaine and Dexmedetomidine); Group R(Ropivacaine Only): Patients' satisfaction were assessed verbally 48 hours after surgery using a 5- point Likert scale (5=completely satisfied, 4=quite satisfied, 3=slightly dissatisfied, 2=dissatisfied, 1=very dissatisfied).
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Number analyzed (Participants) | 30 | 30
Participants
  1 point of 5- point Likert scale | 0 | 0
  2 point of 5- point Likert scale | 0 | 0
  3 point of 5- point Likert scale | 1 | 7
  4 point of 5- point Likert scale | 9 | 17
  5 point of 5- point Likert scale | 20 | 6
Statistical Analysis 1: Comparison: Group RD(Ropivacaine and Dexmedetomidine) vs Group R(Ropivacaine Only); Test type: Other — difference test; Kendall's tau-b correlation coefficient = 0.470

3. Secondary Outcome: Number of Participants With Postoperative Rescue Analgesic Administration
Description: a rescue analgesic morphine 5mg will be administered for any pain score ≥4 （0: no pain--means the minimum value; 10: worst possible pain--means the maximum value)
Time Frame: Hour 24, Hour 48 after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Group RD(Ropivacaine and Dexmedetomidine); Group R(Ropivacaine Only): An extra rescue analgesic morphine 5 mg was given when the NRS was ≥ 4 at rest. The time of the first rescue analgesic requirement and the total morphine consumption in the first 48 hours were recorded.
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Number analyzed (Participants) | 30 | 30
Participants | 1 | 1

4. Secondary Outcome: Adverse Events
Description: including nausea, vomiting, hypotension, bradycardia, and respiratory depression
Time Frame: Hour 48 after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Group RD(Ropivacaine and Dexmedetomidine); Group R(Ropivacaine Only): Postoperative adverse effects such as nausea, vomiting, hypotension, hypoxemia, cardiac arrhythmia and the complications from the drugs and technique (local anesthetic toxicity, vascular puncture) were recorded and treated.
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Number analyzed (Participants) | 30 | 30
Participants | 5 | 3
Statistical Analysis 1: Comparison: Group RD(Ropivacaine and Dexmedetomidine) vs Group R(Ropivacaine Only); Test type: Superiority; p > 0.05, Fisher Exact; Risk Ratio (RR) = 0.64

ADVERSE EVENTS:
Time Frame: Postoperative 48h adverse effects such as nausea, vomiting, hypotension, hypoxemia, cardiac arrhythmia and the complications from the drugs and technique (local anesthetic toxicity, vascular puncture) were recorded and treated.
Arm/Group | Group RD(Ropivacaine and Dexmedetomidine) | Group R(Ropivacaine Only)
Serious Adverse Events (participants affected / at risk) | 3/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group RD(Ropivacaine and Dexmedetomidine) (N=30) | Group R(Ropivacaine Only) (N=30)
bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group RD(Ropivacaine and Dexmedetomidine) (N=30) | Group R(Ropivacaine Only) (N=30)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes